CLINICAL TRIAL: NCT02537704
Title: Translational Study for Overweight and Obesity Management in Adults Using the "Group Lifestyle Balance Program" in Primary Care Clinics and Public Hospitals From Sonora, México
Brief Title: Translational Study for Obesity Management in Mexican Adults Using the "Group Lifestyle Balance Program"
Acronym: GLBOMEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Professor (Full)., Universidad de Sonora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPPMEX-077
Record Dates: First submitted 2015-08-25; First posted 2015-09-02 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Translational; Diabetes Prevention Program; Group Lifestyle Balance Program
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Lifestyle Balance Program (Experimental): Participants will be assigned to an adaptation of the "Group Lifestyle Balance Program", a behavioral curriculum implemented in the Diabetes Prevention Program Study. The Group Lifestyle Balance Program will be provided weekly for the first 3.5 months, bi-weekly from 3.5 to 6 months and then monthly until 12 months. Health care providers will be trained for the implementation of the intervention.
  Additionally, participants will attend at least one monthly visit with a nutritionist (individually).
  The lifestyle objectives for participants will be as follows:
  1. To lose 5-10% of initial weight through healthy eating.
  2. To do 150 minutes of physical activity each week.
  Interventions: Behavioral: Group Lifestyle Balance Program

INTERVENTIONS:
Behavioral: Group Lifestyle Balance Program

SUMMARY:
Obesity is the main modifiable risk factor for the development of chronic diseases in Mexico. Several randomized controlled trials have shown that intensive lifestyle programs are efficacious for the management of obesity. These programs include frequent sessions (14 or more contacts in the first 6 months) focused on diet and physical activity and use a behavior change protocol. In Mexico most primary care clinics and public hospitals apply traditional treatments for obesity management, which have limited effect on weight loss. This study would provide scientific evidence for an effective model for obesity management. Objective. The purpose of this study is to evaluate the effectiveness of the "Group Lifestyle Balance Program" for overweight and obesity management in adults, in primary care clinics and public hospitals from Sonora. This is a translational clinical study. Healthcare providers from the participating clinics will be trained with the Group Lifestyle Balance Program before its implementation. The primary outcome measurement is the change in body weight from baseline to 6 months and 12 months. Changes in body mass index, waist circumference, systolic and diastolic blood pressure, depression, quality of life and stress scales will be measured in patients receiving the program before and 6 and 12 months after starting the program. Additionally, biochemical parameters (fasting glucose, total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, fasting insulin, Homeostatic Model Assessment- Insulin Resistance (HOMA-IR) and liver enzymes [Aspartate transaminase (AST), Alanine Aminotransferase (ALT)] will be evaluated from baseline to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age and <65)
* Overweight or Obese (BMI >25 kg/m2 y <50 kg/m2)
* Availability and motivation to attend the intervention program
* Patients who would benefit from participating in the program according to the health providers
* Signing an informed consent

Exclusion Criteria:

* Medical conditions affecting body weight significantly
* Pregnancy or nursing
* Bariatric surgery
* Being unable to participate in regular moderate physical activity
* Blood pressure >160 mm/Hg
* HbA1c>9

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Change in body weight from baseline to 6 months and change in body weight from baseline to 12 months

SECONDARY OUTCOMES:
Change in waist circumference | Change in waist circumference from baseline to 6 months and change in waist circumference from baseline to 12 months
Change in body fat percentage | Change in body fat percentage from baseline to 6 months and change in body fat percentage from baseline to 12 months
Change in the Beck Depression Inventory score | Change in the Beck Depression Inventory score from baseline to 6 months and change in in the Beck Depression Inventory score from baseline to 12 months
Change in the Short Form-36 Health Survey score | Change in the Short Form-36 Health Survey score from baseline to 6 months and change in the SF-36 Health Survey score from baseline to 12 months
Change in the Perceived Stress Scale (PSS) -14 score | Change in the Perceived Stress Scale (PSS) -14 score from baseline to 6 months and change in the Perceived Stress Scale PSS-14 score from baseline to 12 months
Change in systolic and diastolic blood pressure | Change in systolic and diastolic blood pressure from baseline to 6 months and change in systolic and diastolic blood pressure from baseline to 12 months
Change in fasting glucose | Change in fasting glucose from baseline to 12 months
Change in total cholesterol | Change in total colesterol from baseline to 12 months
Change in LDL-cholesterol | Change in LDL-cholesterol from baseline to 12 months
Change in HDL-cholesterol | Change in HDL-cholesterol from baseline to 12 months
Change in triglycerides | Change in triglycerides from baseline to 12 months
Change in fasting insulin | Change in fasting insulin from baseline to 12 months
Change in HOMA-IR | Change in HOMA-IR from baseline to 12 months
Change in liver enzymes [AST and ALT] | Change in liver enzymes [AST and ALT] from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolando G Díaz, Ph.D., Principal Investigator — Universidad de Sonora
Locations (5):
- Mexico (5):
  - Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora
  - Centro de Salud Urbano Dr. Domingo Olivares, Hermosillo, Sonora
  - Hospital General del Estado de Sonora, Hermosillo, Sonora
  - Hospital Ignacio Chávez, Hermosillo, Sonora
  - Centro Avanzado de Atención a la Salud (CAAPS), Hermosillo, Sonora

REFERENCES:
- [Derived] Ruelas AL, Martinez Contreras TJ, Esparza Romero J, Diaz Zavala RG, Candia Plata MDC, Hingle M, Armenta Guirado B, Haby MM. Factors influencing adults to drop out of intensive lifestyle interventions for weight loss. Transl Behav Med. 2023 Apr 15;13(4):245-254. doi: 10.1093/tbm/ibac112. PMID 36694376